CLINICAL TRIAL: NCT04383197
Title: Effects of 12 Weeks of Endurance Exercise Training Alone or in Combination With Glucagon Like Peptide 1 Receptor Agonist (GLP-1 RA) Treatment on Insulin Secretory Capacity in Type 2 Diabetes
Brief Title: Exercise and GLP-1 RA on Insulin Secretion
Acronym: EXISECRET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Flemming Dela, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-19008233
Record Dates: First submitted 2020-05-04; First posted 2020-05-12 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes
Keywords: Insulin secretion; Beta cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Semaglutide treatment (Experimental): 3 months of therapeutic semaglutide treatment
  Interventions: Drug: Semaglutide
- Semaglutide and Endurance exercise (Experimental): 12 weeks of endurance exercise concomitant to semaglutide treatment
  Interventions: Behavioral: Endurance exercise training; Drug: Semaglutide
- Endurance exercise (Experimental): 12 weeks of endurance exercise
  Interventions: Behavioral: Endurance exercise training

INTERVENTIONS:
Behavioral: Endurance exercise training — Ergometer cycling at 70 % of VO2 max, 45 minutes, 3 times a week
  Arms: Endurance exercise; Semaglutide and Endurance exercise
Drug: Semaglutide — 3 months of therapeutic treatment with semaglutide
  Arms: Semaglutide and Endurance exercise; Semaglutide treatment

SUMMARY:
The purpose of this study is to determine the effect of endurance exercise on insulin secretory capacity, alone or in addition to treatment with the glucagon-like-peptide receptor agonist semaglutide, in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The effects of endurance exercise alone or in addition to treatment with glucagon-like- peptide receptor agonists on insulin secretory capacity, will be determined in patients with type 2 diabetes.

Included patients will be randomized to either 12 weeks of endurance exercise training 3 times a week or therapeutical treatment with semaglutide for 3 months followed by 12 weeks of endurance exercise training 3 times a week. Insulin secretory capacity will be determined by hyperglycemic clamp method before and after.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* BMI 28-35
* Moderately preserved insulin secretory capacity (determined by glucagon test)

Exclusion Criteria:

* Insulin treatment
* Hypertension grade 3
* Heart disease
* Medical history with pancreatitis
* Diagnosed with neuropathy
* Excessive alcohol consumption
* Any condition that would interfere with the protocol.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Insulin secretion | Change from baseline insulin secretion after Exercise intervention(12 weeks).
  By hyperglycemic clamp
Insulin secretion | Change from baseline insulin secretion after 3 months of therapeutic semaglutide treatment
  By hyperglycemic clamp
Insulin secretion | Change from baseline insulin secretion after 3 months of combined exercise and therapeutic semaglutide treatment
  By hyperglycemic clamp

SECONDARY OUTCOMES:
Insulin secretion | Before and after (3 days) Exercise intervention (12 weeks). Before and after 3 months of therapeutic semaglutide treatment
  By Oral glucose tolerance test
insulin sensitivity | Before and after (2 days) Exercise intervention(12 weeks). Before and after 3 months of therapeutic semaglutide treatment
  Derived from hyperglycemic clamp and HOMA-IR
Changes in plasma bone markers | Before and after (2 days) Exercise intervention (12 weeks). Before and after 3 months of therapeutic semaglutide treatment
  Changes in baseline CTX, PNIP, Osteocalcin and alkaline phosphatase
Glucose homeostasis | Before and after (2 days) Exercise intervention (12 weeks). Before and after 3 months of therapeutic semaglutide treatment
  Changes in HbA1c
Cardiorespiratory fitness | Before and after (3 days) Exercise intervention (12 weeks). Before and after 3 months of therapeutic semaglutide treatment
  Changes in maximal oxygen uptake
Body composition | Before and after (3 days) Exercise intervention (12 weeks). Before and after 3 months of therapeutic semaglutide treatment
  By DXA

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Dela, Principal Investigator — University of Copenhagen
Locations (1):
- Xlab, Center for Healthy Aging, Department of Biomedical Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Can be provided upon reasonable request

REFERENCES:
- [Derived] Ingersen A, Schmucker M, Alexandersen C, Graungaard B, Thorngreen T, Borch J, Holst JJ, Helge JW, Dela F. Effects of Aerobic Training and Semaglutide Treatment on Pancreatic beta-Cell Secretory Function in Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2023 Oct 18;108(11):2798-2811. doi: 10.1210/clinem/dgad326. PMID 37265222